CLINICAL TRIAL: NCT00024076
Title: Radiofrequency Ablation of Pulmonary Malignancy
Brief Title: Radiofrequency Ablation in Treating Patients With Refractory or Advanced Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068889; UCLA-9908024; NCI-G01-2011
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Lung Cancer; Malignant Mesothelioma; Metastatic Cancer; Thymoma and Thymic Carcinoma
Keywords: recurrent non-small cell lung cancer; recurrent small cell lung cancer; recurrent malignant mesothelioma; recurrent thymoma and thymic carcinoma; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; pulmonary carcinoid tumor; lung metastases
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma, Malignant; Neoplasm Metastasis; Thymoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Radiofrequency ablation uses high-frequency electric current to kill tumor cells. CT-guided radiofrequency ablation may be effective treatment for lung cancer.

PURPOSE: Phase II trial to study the effectiveness of radiofrequency ablation in treating patients who have refractory or advanced lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of radiofrequency ablation in patients with refractory or advanced pulmonary malignancies.
* Determine the efficacy of this treatment, in terms of local control, in these patients.
* Determine whether CT scan is a reasonable imaging assessment tool for treatment delivery and follow-up in these patients.

OUTLINE: Patients undergo percutaneous CT-guided radiofrequency ablation directly to the tumor over 2 hours.

Patients are followed at 1, 3, 6, and 12 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a primary or secondary intrathoracic malignancy

  * Any cell type or origin
  * Involving the intrapulmonary, mediastinal, or pleural/chest wall
  * Inoperable primary or metastatic cancer to the lung
* Refractory to or not amenable to conventional therapy (e.g., surgery, chemotherapy, or radiotherapy)
* Single or multiple lesions that are non-contiguous with vital structures or organs such as:
* Trachea
* Heart
* Aorta
* Great vessels
* Esophagus
* Less than 5 cm in largest dimension
* Accessible via percutaneous transthoracic route
* Hepatic:

  * Coagulation profile normal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-05; Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Suh, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States